CLINICAL TRIAL: NCT03685903
Title: Prospective Observational Study for the Detection of Duodenal Papilla Using Capsule Endoscopy and Comparison of Images With EUS/ERCP Procedure in Pancreaticobiliary and Periampullary Pathology
Brief Title: Study for the Detection of Duodenal Papilla Using Capsule Endoscopy and Comparison of Images With EUS/ERCP Procedure.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Capso Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CLN-CVI-4801
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Patients Indicated for Periampullary or Pancreaticobiliary Examination
MeSH Terms: interventions — Capsule Endoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CapsoCam® Plus (SV-3) capsule endoscope (Experimental): Endoscope Capsule
  Interventions: Device: CapsoCam® Plus (SV-3) capsule endoscope

INTERVENTIONS:
Device: CapsoCam® Plus (SV-3) capsule endoscope — Endoscope Capsule

SUMMARY:
This observational Non-Significant Risk (NSR) Study will be used to assess the ability of CapsoCam® Plus (SV-3) capsule endoscope to detect the duodenal papilla and visualize pathology or abnormalities in the periampullary area and will prospectively compare the capsule endoscopy and EUS/ERCP pictorial images acquired in procedures conducted in a minimum of 20 and a maximum of 200 research patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age.
* Provided written HIPAA Informed Consent in the IRB approved language.
* Patients indicated for periampullary or pancreaticobiliary examination, with prior cross-sectional imaging (CT/MRI/US/other) performed within past 6 months.

Exclusion Criteria:

* Patients with existing biliary stent will be excluded
* EUS/ERCP exclusion criteria: per medical practice, including:

  1. Patient refusal to undergo procedure, unstable cardiopulmonary, neurologic, or cardiovascular status; existing bowel perforation
  2. Structural abnormalities of esophagus, stomach, small intestine at the discretion of physician.
* Capsule Endoscopy (CE) exclusion criteria:

  1. CE exclusion criteria: difficulty swallowing, pregnancy, known motility issues (gastroparesis), known strictures, gastrointestinal obstructions, fistula or significantly distorted anatomy.
  2. Medical history of receipt of surgery, oncologic therapy, or radiation therapy who, in the opinion of the investigator, are at greater risk of capsule endoscope retention.
  3. Any other contra-indicated condition as noted on the CapsoCam® Plus (SV-3) Instructions for Use, package insert.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
The ability to detect and visualize the duodenal papilla | during capsule endoscopy procedure
  Rate of duodenal papilla detection

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No